CLINICAL TRIAL: NCT02574923
Title: Outcomes of Autologous Bone Marrow Mononuclear Cells for Cerebral Palsy: A Self-Controlled Clinical Trial
Brief Title: Outcomes of Stem Cells for Cerebral Palsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vinmec Healthcare System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBG 002
Record Dates: First submitted 2015-10-09; First posted 2015-10-14 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Stem Cells
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stem cell transplantation (Experimental): 2 intrathecal administrations of autologous bone marrow mononuclear cells at baseline and 3 months afterward
  Interventions: Biological: Autologous Bone Marrow Mononuclear Cells

INTERVENTIONS:
Biological: Autologous Bone Marrow Mononuclear Cells — Transplantation of Autologous Bone Marrow Mononuclear Cells

SUMMARY:
The aim of this study is to assess the safety and effectiveness of autologous bone marrow mononuclear stem cells in patients with cerebral palsy.

DETAILED DESCRIPTION:
The aim of this study is to assess the safety and effectiveness of autologous bone marrow mononuclear stem cells in 30 patients with cerebral palsy at Vinmec International Hospital, Hanoi, Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy of any types caused by oxygen deprivation.

Exclusion Criteria:

* Epilepsy
* Hydrocephalus with ventricular drain
* Coagulation disorders
* Allergy to anesthetic agents
* Severe health conditions such as cancer, failure of heart, lung, liver or kidney
* Active infections

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Total Score of Gross Motor Function Measure (GMFM)-88 | 3 months and 6 months after transplantation
  GMFM-88
Change in Gross Motor Function Measure (GMFM)-66 Percentile | 3 months and 6 months after transplantation
  GMFM-66 percentile

SECONDARY OUTCOMES:
Change in Muscle tone | 3 months and 6 months after transplantation
  Muscle tone are assessed by Modified Ashworth Scale
Number of adverse events | Through study completion, an average of 6 months
  Examples of adverse events to look for: anaphylaxis, allergy, respiratory distress, fever, infections, vomit, epilepsy
Change in Denver Developmental Score | 3 months and 6 months after transplantation
  Denver II
Change in Quality of Life | 3 months and 6 months after transplantation
  Quality of life questionnaire for cerebral palsy (CPQOL)

CONTACTS AND LOCATIONS:
Overall Officials: Liem T Nguyen, MD., PhD., Study Chair — Vinmec Healthcare System
Locations (1):
- Vinmec International Hospital, Hanoi, Vietnam

REFERENCES:
- [Background] Sharma A, Sane H, Gokulchandran N, Kulkarni P, Gandhi S, Sundaram J, Paranjape A, Shetty A, Bhagwanani K, Biju H, Badhe P. A clinical study of autologous bone marrow mononuclear cells for cerebral palsy patients: a new frontier. Stem Cells Int. 2015;2015:905874. doi: 10.1155/2015/905874. Epub 2015 Feb 18. PMID 25788947
- [Derived] Than UTT, Nguyen LT, Nguyen PH, Nguyen XH, Trinh DP, Hoang DH, Nguyen PAT, Dang VD. Inflammatory mediators drive neuroinflammation in autism spectrum disorder and cerebral palsy. Sci Rep. 2023 Dec 18;13(1):22587. doi: 10.1038/s41598-023-49902-8. PMID 38114596
- [Derived] Nguyen TL, Nguyen HP, Nguyen TK. The effects of bone marrow mononuclear cell transplantation on the quality of life of children with cerebral palsy. Health Qual Life Outcomes. 2018 Aug 14;16(1):164. doi: 10.1186/s12955-018-0992-x. PMID 30107811